CLINICAL TRIAL: NCT00961077
Title: A Prospective Phase II Study of Attenuated S-1 and Oxaliplatin(Attenuated SOX) as First-line Treatment in Elderly Patients With Relapsed or Metastatic Gastric Cancer
Brief Title: Attenuated SOX as First-line Treatment in Elderly Patients With Relapsed or Metastatic Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Jong-Ho Won, Soonchunhyang University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCH-HO-GC-01
Record Dates: First submitted 2009-08-17; First posted 2009-08-18 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Elderly; S-1; Oxaliplatin; First-Line; Gastric Cancer
Keywords: elderly; S-1; Oxaliplatin; relapsed or metastatic gastric cancer
MeSH Terms: conditions — Stomach Neoplasms; Recurrence | interventions — S 1 (combination); titanium silicide; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: S-1 (TS-1) and Oxaliplatin (Oxalitin) — S-1(TS-1) 60mg/m2/day (D1-14) Oxaliplatin: 85mg/m2 + 5DW 250mL MIV over 2-hours
  every 3 weeks

SUMMARY:
Stomach cancer is the most common malignant disease and the second most common cause of cancer-related deaths in the Korea. The elderly are primarily affected by the disease with most gastric cancer-related deaths occuring in patients aged 65 years or older. Systemic chemotherapy improves the quantity and quality of life in patients with gastric cancer when compared with best supportive care. However, elderly cancer patients often present with concomitant co-morbidities and age-associated physiologic problems that make the selection of optimal treatment difficult. There is also uncertainty about the use of systemic palliative chemotherapy in elderly patients because of under representation of this age group in clinical trials. Therefore, this phase II trial was planned to investigate efficacy and toxicities of combination chemotherapy with attenuated dose of S-1 and oxaliplatin (attenuated SOX)in patients with elderly AGC

DETAILED DESCRIPTION:
Treatment scheme

* S-1 60mg/m2/day (D1-14) Oxaliplatin: 85mg/m2 + 5DW 250mL MIV over 2-hours

Each cycle is repeated every 3 weeks

Response evaluation will be performed every 2 cycles

Repeated cycles of treatment will be given for this study unless there is confirmed disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age : more than 70 to 80 and ECOG PS 0-2
* Age : more than 65 to less than 70 and ECOG PS 2
* Histological or pathologically confirmed adenocarinoma
* Relapsed or metastatic adenocarcinoma of stomach
* No previous chemotherapy except adjuvant chemotherapy completed at least 12 months before enrollment
* At least more than one measurable lesion on RECIST criteria
* No radiation history for the target lesion
* An estimated life expectancy of more than 3 months
* Ability for adequate oral intake
* Adequate BM function: defined as WBC≥4000/μL, ANC ≥1500/μL, PLT≥100,000/μL.
* Adequate renal function: defined as Creatinine <1.5mg/dL.
* Adequate hepatic function: defined as total bilirubin < 2.0mg/dL, SGOT/SGPT < normal x 3.
* Written informed consent

Exclusion Criteria:

* Symptomatic brain metastasis or meningeal metastasis.
* Double primary cancer
* Medical history of other cancer within 5 years
* G-I bleeding or intestinal obstruction (other condition that can't have the oral intake)
* Hypersensitivity to the 5-FU or oxaliplatin
* Active infectious disease that need to treat systemically
* Serious medical or psychologic condition: newly developed AMI ( within 6Ms)…

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-08 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
To evaluate response rate of attenuated SOX as first-line chemotherapy in elderly patients with relapsed or metastatic AGC | every 2 cycles

SECONDARY OUTCOMES:
To evaluate progression free survival, overall survival, and toxicities of aSOX-regimen | every 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Cheol Lee, M.D., Principal Investigator — Soonchunhyang University Hospital